CLINICAL TRIAL: NCT02161393
Title: PhysicaL actIvity interVention vErsus puLmonarY Rehabilitation in COPD: The LIVELY COPD Project.
Brief Title: Physical Activity Versus Pulmonary Rehabilitation in COPD
Acronym: LIVELY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Western Health and Social Care Trust (Other); Queen's University, Belfast (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Brenda O'Neill, Senior Lecturer in Physiotherapy, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WT12/20
Record Dates: First submitted 2013-05-28; First posted 2014-06-11 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Physical Activity; Pulmonary Rehabilitation; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Activity Intervention (Experimental): 12 week home-based walking programme consisting of weekly physical activity consultations and a pedometer-driven walking programme
  Interventions: Behavioral: Physical Activity Intervention
- Pulmonary Rehabilitation Programme (Active Comparator): 6-week supervised outpatient programme consisting of twice-weekly exercise sessions and once-weekly education sessions.
  Interventions: Behavioral: Pulmonary Rehabilitation Programme

INTERVENTIONS:
Behavioral: Physical Activity Intervention — The 12 week home-based pedometer-driven walking programme will consist of weekly physical activity consultations. Pedometers will be used to set weekly step goals and motivate patients. Patients will wear the pedometer for 7 days and will record their daily steps in a step diary. At the next appointment the step target for the subsequent week will be agreed between the physiotherapist/researcher and participant. Each week thereafter the physiotherapist/researcher and patient will discuss their progress, document their mean daily step count for the previous week, and agree to a new daily step target for the subsequent week. The walking programme will be tailored to the individual and progressed on a weekly basis.
  Arms: Physical Activity Intervention
Behavioral: Pulmonary Rehabilitation Programme — This will be a 6-week supervised outpatient programme. The exercise component will last for one hour and be delivered twice weekly. It will consist of cardiovascular exercises and lower and upper body strengthening exercises. Education sessions will be delivered once weekly. Each patient will be provided with a home exercise programme to complete unsupervised once weekly.
  Arms: Pulmonary Rehabilitation Programme

SUMMARY:
The primary aim of this study is to assess the feasibility of conducting a trial to investigate the effectiveness of a physical activity intervention (physical activity consultation and a pedometer-based walking programme) versus pulmonary rehabilitation in improving physical activity in COPD.

Objectives are:

(i) to assess the feasibility (patient recruitment, adherence, drop-outs and adverse events) of delivering a physical activity intervention in the COPD patient population versus pulmonary rehabilitation; (ii) to explore users perceptions relating to satisfaction and benefits of a physical activity intervention versus pulmonary rehabilitation; (iii) to investigate between and within group change in physical activity, exercise capacity, quality of life, self-efficacy and changes in the transtheoretical model with the physical activity intervention versus pulmonary rehabilitation; and (iv) to examine the cost of delivering a physical activity intervention versus pulmonary rehabilitation for patients with COPD.

The hypothesis for this study is that it will be feasible to conduct a trial that will investigate the effectiveness of a physical activity intervention (physical activity consultation and a pedometer-based walking programme) compared to pulmonary rehabilitation for improving physical activity in COPD. The study will provide important information about interventions designed to promote and maintain physical activity, improve patient outcomes and increase patients' choice relating to exercise and physical activity interventions. It will provide a rationale and data for an adequately powered clinical trial evaluating the effects of a physical activity intervention.

DETAILED DESCRIPTION:
A survey of pulmonary rehabilitation programmes mirrored the results of other UK studies and highlighted that there are not enough programmes available; currently in the UK less than 1.5% of patients with COPD receive pulmonary rehabilitation per year. Only a proportion of patients are targeted i.e. those with moderate to severe disease. The majority of programmes are outpatient-based and are supervised by clinicians. This structured and supervised format of pulmonary rehabilitation does not meet the needs of all patients with high numbers of dropouts and non-adherence; yet alternative options for increasing physical activity for patients with COPD currently do not seem to be offered.

A home-based pedometer-driven walking intervention offers an alternative method of delivering physical activity training that could be provided to larger numbers of patients, at a lower cost and with flexibility around life commitments. It would also provide patients with more choice when deciding whether to participate in exercise or physical activity.

To date no study has compared a home-based walking intervention to structured, supervised pulmonary rehabilitation or the patient preferences or cost of the two programmes. For this reason, there is a need to compare a home-based-walking intervention to the standard method of providing patients with physical activity training, i.e. pulmonary rehabilitation. Therefore this study is essential as it will assess the feasibility of conducting a trial to investigate the efficacy of a physical activity intervention (physical activity consultation and a pedometer-based walking programme) versus pulmonary rehabilitation in improving physical activity in COPD.

ELIGIBILITY:
Inclusion Criteria:

1. The Patient must be referred to pulmonary rehabilitation.
2. The Patient must have a Primary diagnosis of COPD
3. The Patient must have a good understanding of written English (as reported by the individual patient)
4. The Patient must be in a stable phase (not on antibiotics at the time of assessment with the ISWT), and deemed clinically stable by the clinical pulmonary rehabilitation team.

Exclusion Criteria:

1. The inability to safely take part in a walking programme or pulmonary rehabilitation (e.g. unstable angina, neurological, spinal or skeletal dysfunction affecting ability to exercise)
2. The inability to comprehend or follow instructions (e.g. dementia).
3. Clinically unstable (Pulmonary exacerbation or any change in symptoms and medication in the last 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity will be assessed using step counts recorded with an Actigraph activity monitor. | Baseline and at 6-weeks for PR group and 12-weeks for PA group
  The activity monitor is worn for 7 consecutive full days prior to the intervention, and 7 full days immediately after the intervention.

SECONDARY OUTCOMES:
Change from baseline in time spent in physical activity and in sitting using the International Physical Activity Questionnaire | Baseline and at 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
Change from baseline in exercise Capacity using the Incremental Shuttle Walk Test | Baseline, and at 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
Change from baseline in Quality of Life using the EuroQOL-5D | Baseline, and at 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
Change from baseline in Quality of Life using the COPD Assessment Test | Baseline, and at 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
Stage of change in terms of physical activity using the Stages of Change Questionnaire | Baseline, and at 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
  The Stages of Change Questionnaire is the temporal part of the transtheoretical model. It will be used to determine the current stage of change the participant is at in terms of their physical activity behaviour.
Confidence to undertake physical activity using Marcus's Self-Efficacy Questionnaire | Baseline and at 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
  Marcus's Self-Efficacy Questionnaire is a component of the transtheoretical model which will provide more detailed information on each individual's confidence to undertake physical activity in different situations.
Patients' perceptions of both interventions will be obtained via semi-structured interviews. | At 6-weeks for PR group and 12-weeks for PA group
  Information will be collected with regards patient satisfaction with their exercise/activity, information regarding ease of execution, safety and tolerability of the programmes and the outcome measures, views about continuing exercise and suggestions for improving the programmes.
Feasibility of the interventions | End of study
  For both interventions information will be collected on recruitment and retention, dropouts, adherence and adverse events which will be necessary to establish feasibility.
Global Rating of Change Questionnaire | At 6-weeks for PR group and 12-weeks for PA group, and follow up at 18 (PR group) and 24 (PA group) weeks post randomisation
  This is a numerical rating scale about their patient's perception of any change in their physical activity
Physical activity will be assessed using step counts recorded with an Actigraph activity monitor. | At 18 (PR group) and 24 (PA group) weeks post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Brenda O'Neill, PhD, Principal Investigator — University of Ulster
Locations (2):
- United Kingdom (2):
  - Belfast Health and Social Care Trust, Belfast, Co Antrim
  - Western Health and Social Care Trust, Enniskillen